CLINICAL TRIAL: NCT07240844
Title: Enavogliflozin for the Management of Patients With Amyloid CardiomyopaThy - A Randomized, Double-Blind, Placebo-Controlled, Crossover, Multicenter Trial
Brief Title: Enavogliflozin for the Management of Patients With Amyloid CardiomyopaThy
Acronym: EMPACT
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Seoul St. Mary's Hospital (Other)
Collaborators: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Jong-Chan Youn, MD, PhD, Professor, Seoul St. Mary's Hospital
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: EMPACT; KC25MIDV0449 (Other: Seoul St. Mary's Hospital, The Catholic University of Korea)
Record Dates: First submitted 2025-09-28; First posted 2025-11-21 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-08

CONDITIONS: Amyloid Cardiomyopathy
Keywords: Amyloid Cardiomyopathy; Enavogliflozin; Sodium-Glucose Cotransporter 2 Inhibitor
MeSH Terms: conditions — Amyloid Neuropathies, Familial | interventions — Enavogliflozin

STUDY DESIGN:
Intervention Model Description: Prospective, multi-center, double-blind, randomized controlled, crossover, superiority trial
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Enavogliflozin (Experimental): Administer Enavogliflozin 0.3 mg
  Interventions: Drug: Enavogliflozin 0.3mg
- Placebo (Placebo Comparator): Administer placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Enavogliflozin 0.3mg — Participants will receive Enavogliflozin 0.3 mg orally once daily for 12 weeks. The drug is administered in tablet form and is taken during the first or second treatment period of a crossover design.
  Arms: Enavogliflozin
Drug: Placebo — Participants will receive placebo orally once daily for 12 weeks. The drug is administered in tablet form and is taken during the first or second treatment period of a crossover design.
  Arms: Placebo

SUMMARY:
This study aims to evaluate the safety and effectiveness of Enavogliflozin 0.3 mg, an SGLT2 inhibitor, in patients with amyloid cardiomyopathy. Participants will take both the study drug and a placebo in two separate periods, with a wash-out period in between. The goal is to determine whether Enavogliflozin is safe and effective for treating amyloid cardiomyopathy.

DETAILED DESCRIPTION:
Patients with a confirmed diagnosis of cardiac amyloidosis and symptomatic heart failure (NYHA class II-III) will be recruited.

Participants will be randomized to receive either the study drug or placebo and will undergo baseline and 12-week assessments, including the Kansas City Cardiomyopathy Questionnaire (KCCQ), 6-minute walk test, and cardiopulmonary exercise testing. Following a 4-week washout period, participants will cross over to the alternate treatment arm (study drug or placebo) and repeat the same assessments at baseline and 12 weeks.

The primary endpoint will be the change in KCCQ Clinical Summary Score (KCCQ-CSS).

ELIGIBILITY:
Inclusion Criteria:

1. Adults aged 19 years or older
2. Diagnosed with amyloid cardiomyopathy confirmed by cardiac biopsy or non-invasive imaging
3. Presence of heart failure symptoms corresponding to NYHA functional class II-III
4. Patients on stable oral diuretic use, without dose changes exceeding 50% of the previous dose, for at least 2 weeks prior to study enrollment
5. Ambulatory (able to walk)
6. Able to provide written informed consent for study participation

Exclusion Criteria:

1. Pregnant or breastfeeding women
2. Active infection
3. Major cardiovascular events (e.g., myocardial infarction, stroke) within the past 6 months
4. Scheduled for coronary revascularization, CRT-D implantation, atrial flutter/fibrillation ablation, or valve surgery
5. History of heart transplantation
6. Estimated glomerular filtration rate (eGFR) < 60 ml/min/1.73 m² (calculated by CKD-EPI formula)
7. No history of cancer within the past 5 years at screening (except borderline cancers without recurrence for 2-3 years; multiple myeloma with cardiac involvement is classified as cardiac amyloidosis and is exempt)
8. Heart failure primarily caused by severe left sided valvular disease or ischemic heart disease (except if valvular disease is corrected)
9. Type 1 diabetes mellitus or insulin-dependent diabetes
10. History of ketoacidosis, complicated urinary or genital infections, or kidney stones
11. Systolic blood pressure < 80 mmHg or symptomatic hypotension
12. Major surgery within 90 days prior to enrollment
13. Known hypersensitivity or allergic reaction to the study drug or its components
14. Moderate to severe liver impairment
15. Chronic alcohol or substance abuse
16. Residing in long-term care facilities (e.g., nursing homes)
17. Unable to understand or comply with study drug, procedures, or follow-up, or who are deemed by the investigator to be unlikely to complete the study

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Estimated)
Dates: Start 2025-11-24 (Estimated); Primary Completion 2027-04-29 (Estimated); Study Completion 2027-05-31 (Estimated)

PRIMARY OUTCOMES:
Change in KCCQ-CSS from baseline to Week 12 | Baseline and Week 12
  Change in the Clinical Summary Score of the Kansas City Cardiomyopathy Questionnaire (KCCQ-CSS) from baseline to 12 weeks after treatment initiation.
  The KCCQ-CSS is a patient-reported outcome measure that assesses symptom frequency and physical limitation in patients with heart failure.
  Scores range from 0 to 100, with higher scores indicating better symptom status and physical function (i.e., better health status).
  A higher change from baseline reflects an improvement in clinical status.

SECONDARY OUTCOMES:
Change in 6-Minute Walk Distance | Baseline and Week 12
  Change in distance walked in 6 minutes from baseline to Week 12. Higher distance indicates better exercise capacity.
Change in log-transformed NT-proBNP levels | Baseline and Week 12
  Change in log-transformed NT-proBNP levels after 12 weeks of treatment compared to baseline
Change in Body Weight | Baseline and Week 12
  Change in body weight in kilograms from baseline to Week 12
Change in Body Fat Percentage | Baseline and Week 12
  Change in body fat percentage from baseline to Week 12
Change in Extracellular Water Ratio | Baseline and Week 12
  Change in the ratio of extracellular water to total body water from baseline to Week 12
Incidence of Worsening Heart Failure Events or Death | From baseline to Week 12 during each treatment period (excluding the 4-week washout period)
  Occurrence of worsening heart failure events (defined as emergency outpatient visit or unplanned hospitalization due to heart failure) or death

OTHER OUTCOMES:
Change in maximal oxygen consumption (VO₂ max) | Baseline and Week 12
  Change in VO₂ max measured by cardiopulmonary exercise testing (CPET) from baseline to Week 12.
  Higher values indicate better cardiorespiratory fitness.

CONTACTS AND LOCATIONS:
Overall Officials: Jong-Chan Youn, MD, PhD, Principal Investigator — Seoul St. Mary's Hospital, The Catholic University of Korea
Locations (2):
- South Korea (2):
  - Samsung Medical Center, Seoul
  - Seoul St. Mary's Hospital, The Catholic University of Korea, Seoul

IPD SHARING:
Plan to Share IPD: Yes
After publication of first manuscript and trial results, the de-identified data will be shared by permission of principle investigator, when asked.
Supporting Information: Study Protocol, CSR
Time Frame: After publication of first manuscript and trial results, the de-identified data will be shared by permission of principle investigator, when asked.
Access Criteria: After publication of first manuscript and trial results, the de-identified data will be shared by permission of principle investigator, when asked.

REFERENCES:
- [Result] Porcari A, Cappelli F, Nitsche C, Tomasoni D, Sinigiani G, Longhi S, Bordignon L, Masri A, Serenelli M, Urey M, Musumeci B, Cipriani A, Canepa M, Badr-Eslam R, Kronberger C, Chimenti C, Zampieri M, Allegro V, Razvi Y, Patel R, Ioannou A, Rauf MU, Petrie A, Whelan C, Emdin M, Metra M, Merlo M, Sinagra G, Hawkins PN, Solomon SD, Gillmore JD, Fontana M. SGLT2 Inhibitor Therapy in Patients With Transthyretin Amyloid Cardiomyopathy. J Am Coll Cardiol. 2024 Jun 18;83(24):2411-2422. doi: 10.1016/j.jacc.2024.03.429. PMID 38866445
- [Result] Packer M, Butler J, Zeller C, Pocock SJ, Brueckmann M, Ferreira JP, Filippatos G, Usman MS, Zannad F, Anker SD. Blinded Withdrawal of Long-Term Randomized Treatment With Empagliflozin or Placebo in Patients With Heart Failure. Circulation. 2023 Sep 26;148(13):1011-1022. doi: 10.1161/CIRCULATIONAHA.123.065748. Epub 2023 Aug 24. PMID 37621153